CLINICAL TRIAL: NCT05543811
Title: The Influence of Food for Special Dietary Use - Spread Enriched With 5-hydroxytryptophan, Theanine and Gamma-aminobutyric Acid on Psychophysiological Functions of Subjects Without Meaningful Organic and Cognitive Disorders
Brief Title: The Influence of Food for Special Dietary Use - Spread Enriched With 5-hydroxytryptophan, Theanine and Gamma-aminobutyric Acid on Psychophysiological Functions of Subjects Without Meaningful Organic and Cognitive Pathology
Acronym: Spread Bogatyr
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal State Budgetary Scientific Institution "Federal Research Centre of Nutrition, Biotechnology (Other)
Collaborators: Group of companies EFKO (Unknown); Russian Science Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 19-76-30014/2022-HV
Record Dates: First submitted 2022-09-13; First posted 2022-09-16 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-04

CONDITIONS: Cognitive Change; Memory; Disturbance, Mild; Emotional Regulation; Concentration Ability Impaired
MeSH Terms: conditions — Lymphoma, Follicular; Emotional Regulation | interventions — Food

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Product for special dietary use (Experimental): Spread Enriched With 5-hydroxytryptophan, Theanine and Gamma-aminobutyric Acid will be given to the subjects enrolled to this arm, 20 gram twice daily with breakfast and supper (instead of butter)
  Interventions: Dietary Supplement: Food for special dietary use
- control (Placebo Comparator): This group will receive standard spread, without theanine, gamma-aminobutyric acid and 5-hydroxytryptophan, twice daily with breakfast and supper with food (instead of butter)
  Interventions: Dietary Supplement: Food for special dietary use

INTERVENTIONS:
Dietary Supplement: Food for special dietary use — Food for special dietary use (spread) with modified ingredients' content will be included to the diet of 70 patients without significant organic pathology for 14 days receiving standard diet, modified by the inclusion of two portions of the spread, 20 grams each for breakfast and dinner

SUMMARY:
This is a single-centre, single-blind, two-arms, controlled study to assess the efficacy and safety of food for special dietary use enriched with 5-hydroxytryptophan, L-theanine and Gamma-aminobutyric acid in generally healthy subjects with no cognitive disturbances

ELIGIBILITY:
Inclusion Criteria:

* willingness to participate;
* age of 18-50 years

Exclusion Criteria:

* pregnancy or breastfeeding;
* significant somatic or psychological disorders

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
change in cognitive function | two weeks
  change in score by Lurie test
change in cognitive function2 | two weeks
  change in Kraepelin&Schulte test score
change in functional status | two weeks
  change in functional status test score
change in anxiety and depression | two weeks
  change in Beck depression inventory score

SECONDARY OUTCOMES:
change in food's taste monotony | two weeks
  change in food's taste monotony

CONTACTS AND LOCATIONS:
Overall Officials: Vasily Isakov, Professor, Study Chair — Federal Research Center of Nutrition and Biotechnology
Locations (1):
- Federal State Budgetary Scientific Institution "Federal Research Centre of Nutrition, Biotechnology, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Yes
Blinded individual participant data may be shared by reasonable request to primary investigator upon study completion
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 2 years after study completion
Access Criteria: reasonable request to primary investigator
URL: http://ion.ru